CLINICAL TRIAL: NCT00469066
Title: Improving the Accuracy of Radiotherapy Planning and Delivery Using Kilovoltage Cone Beam CT Imaging
Brief Title: Cone Beam CT Scanning in Lung and Bladder Cancer.
Status: Completed | Type: Observational
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Cross Cancer Institute (Other)
Responsible Party: Sponsor
Other Study IDs: LU-11-0073
Record Dates: First submitted 2007-05-02; First posted 2007-05-04 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2011-12

CONDITIONS: Lung Neoplasm; Small Cell Carcinoma; Bladder Carcinoma
Keywords: small cell lung cancer; bladder cancer; conformal radiotherapy
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Small Cell; Urinary Bladder Neoplasms; Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
To study changes in tumor and normal organ size and/or position which occur during a course of radiation treatments.

ELIGIBILITY:
Inclusion Criteria:

* Patient has biopsy proven limited stage SCLC
* receiving radical concurrent chemoradiotherapy
* no prior chest RT
* no prior surgical resection of lung tumor
* no prior chemotherapy
* patients' lung tumors should be centrally-located to minimize the effect of respiratory motion
* patient has biopsy proven TCC bladder
* receiving radical concurrent chemoradiotherapy or RT alone
* no prior chemotherapy
* patient signs study-specific consent form

Exclusion Criteria:

* mixed small cell and non small cell histology
* patient not being treated with concurrent chemoradiotherapy
* chemoradiotherapy given sequentially
* previous chest RT
* previous chemotherapy
* prior surgical resection of lung mass
* patient ineligible for pelvic RT
* patient does not sign study consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clniic
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2007-05; Primary Completion 2009-08 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Don Yee, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Cross Cancer Institute, Edmonton, Alberta, Canada